CLINICAL TRIAL: NCT05090111
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Oral Doses of ALG-055009 in Healthy Volunteers and Subjects With Hyperlipidemia, and an Open-Label Assessment of Bioavailability and Food-effect in Healthy Volunteers
Brief Title: A Study of ALG-055009 in Healthy Volunteers and Subjects With Hyperlipidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-055009-301
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALG-055009 (Experimental): Oral dose(s) of ALG-055009 in Healthy Volunteer or subjects with mild hyperlipidemia once daily up to 14 days
  Interventions: Drug: ALG-055009
- Placebo (Placebo Comparator): Oral dose(s) of placebo in Healthy Volunteer or subjects with mild hyperlipidemia once daily up to 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALG-055009 — Single or multiple doses of ALG-055009
  Arms: ALG-055009
Drug: Placebo — Single or multiple doses of Placebo
  Arms: Placebo

SUMMARY:
A Randomized Study of ALG-055009 Drug to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses in Healthy Volunteers and Subjects with Hyperlipidemia

ELIGIBILITY:
Inclusion Criteria for Healthy Subjects:

1. Male and Female between 18 and 55 years old
2. BMI 18.0 to 32.0 kg/m^2

Inclusion Criteria for Subjects with Mild Hyperlipidemia:

1. Male and Female between 18 and 65 years old
2. BMI 18.0 to 35.0 kg/m^2
3. Subject must be on a stable diet for the 3 months prior to screening with a fasting LDL-C level >110 mg/dL at screening

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with Hepatitis A, B, C or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
3. Subjects with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m^2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
4. Subjects with history of thyroid disorder or abnormal thyroid function tests at screening or known sensitivity to thyroid medications
5. Subjects receiving, or urgently requiring, any lipid lowering therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 14 days for Part 1
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 28 days for Part 2
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 35 days for Part 3
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Predose (between -0.25 hours and 0 hours) up to 35 Days
  Pharmacokinetic parameters of ALG-055009 in plasma
Area under the concentration time curve [AUC] | Predose (between -0.25 hours and 0 hours) up to 35 Days
  Pharmacokinetic parameters of ALG-055009 in plasma
Time to maximum plasma concentration [Tmax] | Predose (between -0.25 hours and 0 hours) up to 35 Days
  Pharmacokinetic parameters of ALG-055009 in plasma
Half-life [t1/2] | Predose (between -0.25 hours and 0 hours) up to 35 Days
  Pharmacokinetic parameters of ALG-055009 in plasma
Minimum Plasma Concentration [Cmin] | Predose (between -0.25 hours and 0 hours) up to 35 Days
  Pharmacokinetic parameters of ALG-055009 in plasma
Change in lipid / lipoprotein levels from baseline through Day 28 in Multiple Dose in Subjects with Mild Hyperlipidemia | Screening, Day -1 to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France